CLINICAL TRIAL: NCT02206867
Title: A Randomized, Double-Blind, Parallel-Group Clinical Study to Compare Pharmacokinetics, Safety and Tolerability of LBAL 40 mg With Humira® 40 mg After a Single Subcutaneous Administration in Healthy Male Volunteers
Brief Title: Pharmacokinetics and Safety Study of LBAL in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LG-ALCL001
Record Dates: First submitted 2014-07-30; First posted 2014-08-01 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-06

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- LBAL (Experimental): Developed by LG Life Sciences
  Interventions: Biological: LBAL
- Humira® (Active Comparator): Abbvie
  Interventions: Biological: Humira

INTERVENTIONS:
Biological: LBAL — Anti-inflammatory agents
  Other Names: Adalimumab
  Arms: LBAL
Biological: Humira — Anti-inflammatory agents
  Other Names: Adalimumab
  Arms: Humira®

SUMMARY:
To compare PK, safety and tolerability of LBAL developed by LG Life Sciences Ltd. With those of Humira®.

ELIGIBILITY:
Inclusion Criteria:

1. 20-45 years old healthy males
2. Body mass index 19.0 ~ 28.0 kg/m2

Exclusion Criteria:

1. Diagnosis of current or latent tuberculosis (TB); history of severe active chronic or local infection including TB
2. Severe infection (e.g. sepsis) requiring admission or antibiotics treatment within four weeks prior to administration
3. Clinically relevant previous or concomitant disease including hepatic, renal, neurological, respiratory, gastrointestinal, endocrine, hematologic, oncologic, cardiovascular, urinary, musculoskeletal or psychiatric, autoimmune disease/disorders
4. Chronic or relevant acute infections. A negative result for human immunodeficiency virus (HIV), Hepatitis B (Hep B), and hepatitis C (Hep C) is required for participation (i.e. HIV Ab, HBsAg, HBcAb, HCV Ab)
5. Fever greater than 38.3℃ within a week prior to administration of study drug
6. Previous or current drug abuse

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2014-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in serum over the time interval from 0 extrapolated to infinity | 0 to 65 days
Maximum measured concentration of the analyte in serum | 0 to 65 days

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, M.D., Ph.D., M.B.A, Principal Investigator — Dep. of Clnical Pharmacology, Seoul National University College of Medicine and Hospital